CLINICAL TRIAL: NCT07381634
Title: The Safety and Efficacy of Ondansetron in Reducing Immune Checkpoint Inhibitor-Related Toxicities: A Single-Center Randomized Controlled Clinical Trial
Brief Title: The Safety and Efficacy of Ondansetron in Reducing Immune Checkpoint Inhibitor-Related Toxicities
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Director of Hepatobiliary Surgery, Clinical Professor, Vice President, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2026-021
Record Dates: First submitted 2026-01-03; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma (HCC); IrAE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron Group (Experimental): Standard treatment plan：For patients with hepatocellular carcinoma, the standard treatment plan for liver cancer is adopted, which specifically includes lenvatinib + tislelizumab or lenvatinib + pembrolizumab or atezolizumab + bevacizumab:
  Ondansetron: Maintained at 8mg/qd, orally, until disease progression or intolerance.
  Symptomatic treatments other than 5-HT3 receptor antagonists are permitted, and all concurrent medication situations should be recorded.
  Interventions: Drug: ondansetron
- Control Group (No Intervention): Standard treatment plan：For patients with hepatocellular carcinoma, the standard treatment plan for liver cancer is adopted, which specifically includes lenvatinib + tislelizumab or lenvatinib + pembrolizumab or atezolizumab + bevacizumab
  Symptomatic treatments other than 5-HT3 receptor antagonists are permitted, and all concurrent medication situations should be recorded.

INTERVENTIONS:
Drug: ondansetron — Ondansetron: Maintained at 8mg/qd, orally, until disease progression or intolerance.
  Arms: Ondansetron Group

SUMMARY:
This study is a prospective, randomized, single-center randomized controlled clinical trial to investigate the safety and efficacy of ondansetron in reducing the toxicity associated with immune checkpoint inhibitor treatment. This study plans to enroll 66 patients with hepatocellular carcinoma who are scheduled to receive standard ICI treatment. This study will adopt the 2023 CSCO Guidelines for the Management of Immune checkpoint inhibitor-related toxicity as the main assessment criterion, and take the incidence and severity of irAEs as the main observation indicators to evaluate the effectiveness of ondansetron in reducing the toxicity related to immune checkpoint inhibitor treatment in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 80 years old, both male and female are acceptable.
2. The imaging or pathological diagnosis is hepatocellular carcinoma;
3. It is planned to carry out standard treatment for liver cancer, specifically including lenvatinib + tislelizumab or lenvatinib + pembrolizumab or atezolizumab + bevacizumab.
4. ECOG score: 0 to 2 points;
5. Expected survival period ≥12 weeks;
6. Baseline blood cell count tests and blood biochemistry must meet the following standards:

   White blood cell count ≥3.0×10^9/L; Hemoglobin ≥90 g/L; The absolute neutrophil count is ≥1.5×10^9/L; Platelet count ≥100×10^9/L; Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN). Total bilirubin ≤ twice ULN; Serum creatinine ≤ 1.5 times ULN; Albumin ≥30 g/L;
7. The subjects voluntarily joined this study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. Those who have received treatment with ondansetron within 14 days;
2. Patients with autoimmune diseases;
3. Use of systemic glucocorticoids or other immunosuppressants within 14 days;
4. Those who have previously discontinued ICI treatment due to irAEs;
5. Those with severe liver dysfunction (Child-Pugh grade C);
6. Those with contraindications to ondansetron such as serotonin syndrome or phenylketonuria;
7. Patients allergic to ondansetron;
8. Those who are currently using drugs that may have serious interactions with ondansetron, such as apopmorphine;
9. The researcher evaluated that the patient was unable or unwilling to comply with the requirements of the research protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of irAEs | through study completion, an average of 1 year
  To evaluate whether the prophylactic use of ondansetron can reduce the incidence of immune-related adverse events (irAEs) in patients treated with immune checkpoint inhibitors (ICI). The evaluation criteria mainly refer to the "2023 CSCO Guidelines for the Management of Toxicity Related to Immune Checkpoint Inhibitors", with a focus on the incidence of all grades of irAEs and the incidence of severe irAEs at grade 3 and above. The monitoring scope covers liver and kidney functions, blood routine, cardiac function (electrocardiogram, myocardial injury markers), endocrine function (thyroid function, etc.) and imaging manifestations of pneumonia.
The Severity of irAEs | through study completion, an average of 1 year
  To evaluate whether the prophylactic use of ondansetron can reduce the severity of immune-related adverse events (irAEs) in patients treated with immune checkpoint inhibitors (ICI). The evaluation criteria mainly refer to the "2023 CSCO Guidelines for the Management of Toxicity Related to Immune Checkpoint Inhibitors", with a focus on the incidence of all grades of irAEs and the incidence of severe irAEs at grade 3 and above. The monitoring scope covers liver and kidney functions, blood routine, cardiac function (electrocardiogram, myocardial injury markers), endocrine function (thyroid function, etc.) and imaging manifestations of pneumonia.

SECONDARY OUTCOMES:
ORR | through study completion, an average of 1 year
  Objective Response Rate，according to RECIST v1.1
DCR | through study completion, an average of 1 year
  Disease Control Rate, according to RECIST v1.1

IPD SHARING:
Plan to Share IPD: Yes